CLINICAL TRIAL: NCT00852462
Title: Lung Cancer Symptom Assessment and Management Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Boston Medical Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary E. Cooley, Phd, Nurse Scientist, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 07-404; 5R01CA125256 (NIH)
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Lung Cancer
Keywords: SAMI; Symptom Assessment and Management Intervention Program
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAMI (Experimental): Patients and Health care providers use Symptom Assessment and Management Intervention: patient report symptoms by answering validated questionnaires in a secure online program. The system generates a report for providers that displays symptoms and customized suggestions for their clinical management.
  Interventions: Behavioral: SAMI
- Usual Care (No Intervention): Symptom assessment and management follows customary procedures in each study site.

INTERVENTIONS:
Behavioral: SAMI — Patients and Health care providers use Symptom Assessment and Management Intervention: patient report symptoms by answering validated questionnaires in a secure online program. The system generates a report for providers that displays symptoms and customized suggestions for their clinical management.
  Arms: SAMI

SUMMARY:
The purpose of this study is to develop and test the usability of a computerized symptom assessment and management intervention system in a laboratory setting (phase I) and its feasibility in a clinical setting in a group randomized trial (phase II).

ELIGIBILITY:
Inclusion Criteria:

* HCPs: attending physician, thoracic medical oncologist, expected to work in the setting for at least 2 years.
* Patients: 21 years of age or older; diagnosis of Stage IIIA, IIIB, IV non-small cell lung cancer OR limited or extensive stage small cell lung cancer; receiving care in the out-patient setting; receiving treatment with chemotherapy +/- additional therapies; English speaking.

Exclusion Criteria:

* Patients: Any patient who needs emergent care, routine visits scheduled less than once a month

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2008-05; Primary Completion 2012-08 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
% completion of intervention use and adherence to suggested symptom management strategies. | 2 years

SECONDARY OUTCOMES:
Health-related quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Cooley, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts